CLINICAL TRIAL: NCT02396667
Title: Accuracy of 5D LB Ultrasound in Prediction of Birth Weight in Macrosomic Babies: A Pilot Study
Brief Title: Accuracy of 5D LB Ultrasound in Prediction of Birth Weight in Macrosomic Babies : A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mohamed laban, professor, Ain Shams University
Other Study IDs: m2493
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Macrosomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pregnant women with macrosomia: Pregnant wo.en between 37 and 42 weeks with fetal macrosomia as suspected by clinical estimation and 2D ultrasound.
  Interventions: Other: 5D ultrasound

INTERVENTIONS:
Other: 5D ultrasound — Measure the femur length by 5DLB to calculate fetal weight

SUMMARY:
5D and 2D ultrasounds will be done for pregnant women with macrosomic fetuses to determine estimated fetal weight using hadlock formula. The accuracy of fetal weight obtained by ultrasound will be compared to actual birth weight.

ELIGIBILITY:
Inclusion Criteria:

* 37 to 42 weeks gestation
* macrosomic fetuses
* maternal diabetes

Exclusion Criteria:

* intrauterine fetal death
* multiple pregnancy
* congenital anomaly
* nonvisualized fetal parts

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women between 37 and 42 weeks with macrosomic fetuses.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of 5D ultrasound in predicting actual birth weight in comparison to 2D ultrasound. (estimated by hadlock formula - Accuracy of estimated fetal weight by ultrasound will be compared to actual birth weight) | 72hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt